CLINICAL TRIAL: NCT05685030
Title: Evaluation of the Effectiveness of Probiotic Strains (L. Reuteri CCT 7862) and (B. Lactis CCT 7858 + L. Rhamnosus - CCT 7863) in Reducing Colic and Improving Gastrointestinal Health in Newborn
Brief Title: Probiotics Strains for Infant Colic
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Responsible Party: Principal Investigator, Monique Michels, Principal Investigator, Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 63543922.2.0000.0119
Record Dates: First submitted 2022-12-12; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Colic
Keywords: infant colic; probiotic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Intervention Model Description: Phase II randomized, placebo-controlled, triple-blind clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): product vehicle (sunflower oil)
  Interventions: Dietary Supplement: Placebo
- Limosilactobacillus reuteri CCT 7862 (Experimental): Limosilactobacillus reuteri CCT 7862 - 1 x 10e9 UFC/ daY.
  Interventions: Dietary Supplement: Limosilactobacillus reuteri CCT 7862
- Bifidobacterium lactis CCT 7858 + Lactobacillus rhamnosus CCT 7863 (Experimental): Blend: Bifidobacterium lactis CCT 7858 + Lactobacillus rhamnosus CCT 7863 - 1 x 10e9 UFC/ day.
  Interventions: Dietary Supplement: Bifidobacterium lactis CCT 7858 + Lactobacillus rhamnosus CCT 7863

INTERVENTIONS:
Dietary Supplement: Placebo — product vehicle (sunflower oil)
  Arms: Placebo
Dietary Supplement: Limosilactobacillus reuteri CCT 7862 — Limosilactobacillus reuteri CCT 7862 - 1 x 10e9 UFC/ day.
  Arms: Limosilactobacillus reuteri CCT 7862
Dietary Supplement: Bifidobacterium lactis CCT 7858 + Lactobacillus rhamnosus CCT 7863 — Bifidobacterium lactis CCT 7858 + Lactobacillus rhamnosus CCT 7863 - 1 x 10e9 UFC/ day
  Arms: Bifidobacterium lactis CCT 7858 + Lactobacillus rhamnosus CCT 7863

SUMMARY:
Interest in the use of probiotics as a potential treatment to reduce crying in babies with colic has increased lately. Recent studies have reported that the gut microbiota in infants with colic is characterized by lower proportions of Lactobacilli and Bifidobacteria and higher proportions of opportunistic proteobacteria (such as Escherichia coli, Enterobacter aerogenes and Klebsiella spp.) in comparison with the control babies.

Therefore, based on data in the literature, it is understood that there is evidence of the effectiveness of using probiotics, either alone or in the form of a blend, to alleviate the symptoms of infantile colic.

DETAILED DESCRIPTION:
Infantile colic represents a self-limiting temporary condition, which occurs in about one in five babies in the first few months of life, and is characterized by inconsolable crying and fussiness of unknown cause. Despite its benign nature, infantile colic serves as a significant source of maternal anxiety and depression, impaired family functioning, and the most common reason for seeking medical advice in this age group. Infant colic is also associated with sleep problems in babies.

Parents and caregivers often seek medical attention for colic, including the use of medication, plant fiber, lactase, sucrose solution, hypoallergenic diet, and herbal tea. However, there is no single effective and safe intervention for infantile colic.

Interest in the use of probiotics as a potential treatment to reduce crying in babies with colic has increased lately. Recent studies have reported that the gut microbiota in infants with colic is characterized by lower proportions of Lactobacilli and Bifidobacteria and higher proportions of opportunistic proteobacteria (such as Escherichia coli, Enterobacter aerogenes and Klebsiella spp.) in comparison with the control babies. Thus, several researchers have suggested that probiotics may be useful in treating breastfed babies with colic and reducing crying time.

One study showed that administration of Lactobacillus reuteri DSM 17938 improved colic symptoms, although the effectiveness was only seen in breastfed and not formula fed infants. Another study showed that treatment with a combination of L. casei, L. rhamnosus, Streptococcus thermophilus, B. breve, L. acidophilus, B. infantiles, L. bulgaricus and fructooligosaccharides (FOS) reduced the duration of crying by almost 35 min compared to placebo. Furthermore, other authors has reported a reduced incidence of caregiver-reported colic when infants were supplemented with a combination of B. animalis subsp. lactis BB-12 and an unidentified strain of S. thermophilus, although colic was not formally diagnosed by a physician, which reduced the strength of the studies. A recent study on the same BB-12 strain overcame this deficiency by formally diagnosing colic using Rome-III criteria. However, this study showed that the response rate did not significantly improve over placebo until day 21. On the other hand, one study reported that the use of L. rhamnosus GG (ATCC53103) had no significant effect on crying in babies with colic. In another study, no significant differences were found in crying and irritability between the probiotic and placebo groups when supplemented with L. reuteri ATCC55730 or B. lactis BB-12.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 days ± 3 days.
* Informed consent form signed by parents
* Both gender
* Availability to complete scales daily and answer phone calls and/or text messages.

Exclusion Criteria:

* Birth weight <2500 g;
* current intake of antibiotics, prebiotics, or probiotics by the baby or mother;
* Children with known moderate or severe disease of any system (neural, skeletal, muscular, cutaneous, gastrointestinal, respiratory, genital, urinary, immune),
* parental difficulty in understanding study requirements as judged by physician.

Ages: 17 Days to 23 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of probiotics strains by total daily crying time | Change from baseline at three months
  Efficacy of probiotics strains by total daily crying time (minutes for day) recorded by parents daily
Efficacy of probiotics strains by total daily agitation time | Change from baseline at three months
  Efficacy of probiotics strains by total daily agitation time (minutes for day) recorded by parents daily

SECONDARY OUTCOMES:
Safety and Efficacy of probiotics strains | Change from baseline at three months
  Safety and Efficacy of probiotics strains by baby sleep duration (minutes for day) and and sleep quality through scale recorded by parents daily. This Score use a four-point, Likert-type scale, respondents indicate how frequently they exhibit certain sleep behaviors (0 = "few," 1 = "some- times," 2 = "often," and 3 = "almost always").
Safety and Efficacy of probiotics strains | Change from baseline at three months
  Safety and Efficacy of probiotics strains by daily frequency evacuation and stool consistency (Bristol scale). There are seven types of stools (faeces) according to the Bristol Stool Chart. Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhoea and urgency.

CONTACTS AND LOCATIONS:
Locations (1):
- Monique Michels, Criciúma, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No